CLINICAL TRIAL: NCT05150106
Title: Characterization of Clinical Phenotypes of Laryngeal Dystonia and Voice Tremor
Status: Recruiting | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Kristina Simonyan, Professor of Otolaryngology - Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Other Study IDs: 2021P003143
Record Dates: First submitted 2021-11-27; First posted 2021-12-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Laryngeal Dystonia; Spasmodic Dysphonia; Tremor
MeSH Terms: conditions — Dysphonia; Tremor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Voice and speech measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Laryngeal dystonia: Patients with laryngeal dystonia (or spasmodic dysphonia)
  Interventions: Other: Clinical assessments of laryngeal function
- Voice tremor: Patients with voice tremor (essential or dystonic)
  Interventions: Other: Clinical assessments of laryngeal function
- Healthy controls: Healthy research volunteers
  Interventions: Other: Clinical assessments of laryngeal function

INTERVENTIONS:
Other: Clinical assessments of laryngeal function — Participants will undergo acoustic, aerodynamic, respiratory kinematic, nasoendoscopic, and laryngeal EMG recordings, as well as real-time MRI of the upper airway for comprehensive characterization of shared and distinct features of laryngeal dystonia and voice tremor.

SUMMARY:
The researchers will systematically evaluate current and novel clinical voice assessment tools and measures to elucidate distinct clinical phenotypes of those with laryngeal dystonia and voice tremor.

DETAILED DESCRIPTION:
Focal laryngeal dystonia (LD) is a rare neurological voice disorder that interrupts speaking with the intermittent onset of strained-strangled voice quality or causes voicing to stop or produce sudden breathiness. Those suffering from LD commonly report the onset of symptoms 5 years prior to achieving an accurate diagnosis, despite seeing multiple experts. Voice tremor (VT) is another neurological voice disorder that is perceived by listeners as shaky voice quality. Severe VT can result in voice interruptions that sound similar to LD resulting in misdiagnosis by experts. Recent research shows poor reliability in distinguishing those with LD from other voice disorders, largely due to the reliance on perceptual assessment methods and a wide range of clinical criteria without evidence to guide accurate diagnostic approaches. This is particularly true of VT, a voice disorder without clearly documented clinical features such that classification is not possible using current movement disorder consensus-based tremor syndrome criteria. Accurate differential diagnosis of LD from VT is essential to effective treatment planning and management as well as for accurate clinical and epidemiologic characterization and classification. The goal of this research is to systematically characterize individuals with LD and VT using currently available and novel clinical tools to determine distinguishing clinical features highly predictive of their correct diagnosis. Clinical phenotypic features will be compared between groups using acoustic, aerodynamic, laryngeal electromyography (EMG), and nasoendoscopy to quantify periodicity and task-specificity of voice patterns. Novel assessment tools and measures will also be used to study body distribution, condition of speech symptoms, and regularity or intermittency/phoneme-specificity of speech structure movement (kinematic) patterns using real-time magnetic resonance imaging and nasoendoscopy recordings during sustained phonation compared to voice- and voiceless-loaded sentences. Computational modeling will be used to assess aerodynamic, laryngeal EMG and speech structure kinematic patterns to simulate patient-specific acoustic output predictive of group membership as VT or LD. Outcomes of this research will significantly advance our clinical and scientific knowledge regarding optimal clinical tools and measures of LD and VT clinical features that result in a precise diagnosis of these neurological speech disorders.

ELIGIBILITY:
Inclusion criteria:

1. Males and females of diverse racial and ethnic backgrounds;
2. Age 18-80 years;
3. Native English speakers;
4. Right-handed;
5. Normal cognitive status;
6. Patients will have laryngeal dystonia or voice tremor;
7. Healthy controls will be healthy individuals without neurological, psychiatric or otolaryngological problems.

Exclusion criteria:

1. Subjects who are incapable of giving informed consent;
2. Pregnant or breastfeeding women until a time when they are no longer pregnant or breastfeeding. All women of childbearing potential will have a urine pregnancy test performed before MRI, which must be negative for participation in the imaging studies;
3. Subjects with a past or present medical history of (a) neurological problems, such as stroke, movement disorders (other than specified LD and VT in the patient groups), brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases; (b) psychiatric problems, such as schizophrenia, bipolar depression, obsessive-compulsive disorder, alcoholism, drug dependence; (c) laryngeal problems, such as vocal fold paralysis, paresis, vocal fold nodules and polyps, carcinoma, chronic laryngitis;
4. Patients with any other form of dystonia;
5. Patients who have dystonia symptoms at rest or have a presence of mirror dystonia;
6. Patients who are not symptomatic due to treatment with botulinum toxin injections into the affected muscles. The duration of positive effects of botulinum toxin varies from patient to patient but lasts, on average, for 3-4 months. All patients will be evaluated to ensure that they are fully symptomatic and are at least 3 months post-injection before participation;
7. To avoid the confounding effect of centrally acting drugs, all study participants will be questioned about any prescribed or over-the-counter medications as part of their initial screening. Those patients who receive medication(s) affecting the central nervous system will be excluded;
8. Patients will be asked whether they have undergone any head or neck surgery, which resulted in changes in regional anatomy or innervation. Because brain or laryngeal surgery may potentially lead to brain structure and function re-organization, all patients with such a history will be excluded;
9. Subjects who have certain tattoos and ferromagnetic objects in their bodies (e.g., implanted stimulators, surgical clips, prosthesis, artificial heart valve) that cannot be removed for MRI studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with laryngeal dystonia Patients with voice tremor Healthy control individuals
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Differences in voice symptoms | 5 years
  Clinical phenotypic features and speech structure kinematics that distinguish between laryngeal dystonia and voice tremor

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Study Director — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear and University of Utah, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No